CLINICAL TRIAL: NCT02298023
Title: Treatment of Tendon Injury Using Allogenic Adipose-derived Mesenchymal Stem Cells: Phase II Double-Blind Placebo-Controlled Randomized Clinical Trials.
Brief Title: Treatment of Tendon Injury Using Allogenic Adipose-derived Mesenchymal Stem Cells (Rotator Cuff Tear)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun Gun Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALLO-ASC_TR
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Results first posted 2021-06-30 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Rotator Cuff Tear
Keywords: adipose derived mesenchymal stem cell; allogeneic stem cell; Rotator cuff tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mesenchymal stem cell group (Experimental): Received allogenic adipose tissue-derived adult mesenchymal stem cells (10million cells) in fibrin glue scaffold.
  Interventions: Biological: allogenic adipose stem cell injection
- Active control (fibrin glue) group (Active Comparator): Received fibrin glue and normal saline.
  Interventions: Biological: fibrin glue/normal saline injection
- Control (normal saline )group (Placebo Comparator): Received only normal saline.
  Interventions: Biological: normal saline injection

INTERVENTIONS:
Biological: allogenic adipose stem cell injection — Intervention will be done with stem cell injection, 0.5cc (Total: 10 million cells), fibrin glue injection 0.5cc and range of motion exercise.
  Other Names: experimental group
  Arms: Mesenchymal stem cell group
Biological: fibrin glue/normal saline injection — Total 1cc of fibin glue and normal saline mixture injection and range of motion exercise
  Other Names: active control group
  Arms: Active control (fibrin glue) group
Biological: normal saline injection — Total 1cc of normal saline injection and range of motion exercise
  Other Names: placebo group
  Arms: Control (normal saline )group

SUMMARY:
Main purpose of this study is to evaluate efficacy of allogenic adipose-derived mesenchymal stem cells in treatment of tendon injury. ALLO-ASC will be administrated to the patients with supraspinatus partial thickness tear by ultrasonographic guided injection.

DETAILED DESCRIPTION:
Injection volume depends on the size of lesion on ultrasound examination. And all injection will be done under ultrasound guidance. Double blind Randomized placebo controlled study will be done with following 3 groups. Each group will have 8 people, so, the total patients will be 24 people.

1. Stem cell treatment group : stem cell 0.5cc (Total: 10 million cells) + Fibrin glue 0.5cc + range of motion exercise
2. Active control (fibrin glue) group : Normal saline 0.5cc + Fibrin glue 0.5cc + range of motion exercise
3. Control (normal saline) group : Normal saline 0.5cc + Normal saline 0.5cc + range of motion exercise

The investigators will compare the efficacy difference with VAS(visual analog scale, primary outcome), ASES(American Shoulder and Elbow Surgeons) Score, UCLA(University of California, Los Angles) Shoulder Score, DASH(The Disabilities of the Arm, Shoulder and Hand) Score and change of tear size compared to the baseline image assessed by MRI. These measurement will be done at 6 and 12 weeks after injections and long-term follow-up will be also planned to 6 months, 12months and 24 months except for the evaluation of the tear size which will be done at baseline, 3 months and 24 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed as rotator cuff tear (supraspinatus partial thickness tear)
* recurrent pain in spite of conservative treatment such as physical therapy, medication, steroid injection
* symptom duration is over 3 months
* supraspinatus partial thickness tear proven ultrasonography and magnetic resonance image(MRI)
* patient that can understand the clinical trials

Exclusion Criteria:

* patient that underwent other injection treatment within 6 weeks
* some associated diseases (adhesive capsulitis, full thickness supraspinatus tear,. arthritis of related joint to the target lesion, muscle weakness or atrophy, innervated by suprascapular nerve, paralysis of related joint to target lesion, proximal humeral fracture, infectious disease, bilateral rotator cuff tear, generalized pain syndrome, radiculopathy, rheumatoid arthritis, impaired sensibility, dementia, history of allergic or hypersensitive reaction to bovine-derived proteins or fibrin glue and contraindication to MRI
* patient that enrolled other clinical trials within 30 days
* history of drug/alcohol addiction, habitual smoker, operation, allergic reaction to fibrin glue, local anesthetics and bovine-derived proteins and severe medical disease.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Gun Chung, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Isaac C, Gharaibeh B, Witt M, Wright VJ, Huard J. Biologic approaches to enhance rotator cuff healing after injury. J Shoulder Elbow Surg. 2012 Feb;21(2):181-90. doi: 10.1016/j.jse.2011.10.004. PMID 22244061
- [Background] Muller SA, Todorov A, Heisterbach PE, Martin I, Majewski M. Tendon healing: an overview of physiology, biology, and pathology of tendon healing and systematic review of state of the art in tendon bioengineering. Knee Surg Sports Traumatol Arthrosc. 2015 Jul;23(7):2097-105. doi: 10.1007/s00167-013-2680-z. Epub 2013 Sep 21. PMID 24057354
- [Background] Tashjian RZ. Epidemiology, natural history, and indications for treatment of rotator cuff tears. Clin Sports Med. 2012 Oct;31(4):589-604. doi: 10.1016/j.csm.2012.07.001. Epub 2012 Aug 30. PMID 23040548
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] Sanchez M, Azofra J, Anitua E, Andia I, Padilla S, Santisteban J, Mujika I. Plasma rich in growth factors to treat an articular cartilage avulsion: a case report. Med Sci Sports Exerc. 2003 Oct;35(10):1648-52. doi: 10.1249/01.MSS.0000089344.44434.50. PMID 14523300
- [Background] Price R, Sinclair H, Heinrich I, Gibson T. Local injection treatment of tennis elbow--hydrocortisone, triamcinolone and lignocaine compared. Br J Rheumatol. 1991 Feb;30(1):39-44. doi: 10.1093/rheumatology/30.1.39. PMID 1991216
- [Background] Solveborn SA, Buch F, Mallmin H, Adalberth G. Cortisone injection with anesthetic additives for radial epicondylalgia (tennis elbow). Clin Orthop Relat Res. 1995 Jul;(316):99-105. PMID 7634730
- [Background] Johnson GW, Cadwallader K, Scheffel SB, Epperly TD. Treatment of lateral epicondylitis. Am Fam Physician. 2007 Sep 15;76(6):843-8. PMID 17910298
- [Background] Maffulli N, Longo UG, Denaro V. Novel approaches for the management of tendinopathy. J Bone Joint Surg Am. 2010 Nov 3;92(15):2604-13. doi: 10.2106/JBJS.I.01744. PMID 21048180
- [Background] Arce G, Bak K, Bain G, Calvo E, Ejnisman B, Di Giacomo G, Gutierrez V, Guttmann D, Itoi E, Ben Kibler W, Ludvigsen T, Mazzocca A, de Castro Pochini A, Savoie F 3rd, Sugaya H, Uribe J, Vergara F, Willems J, Yoo YS, McNeil JW 2nd, Provencher MT. Management of disorders of the rotator cuff: proceedings of the ISAKOS upper extremity committee consensus meeting. Arthroscopy. 2013 Nov;29(11):1840-50. doi: 10.1016/j.arthro.2013.07.265. Epub 2013 Sep 13. PMID 24041864
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Background] Kon E, Filardo G, Delcogliano M, Presti ML, Russo A, Bondi A, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma: new clinical application: a pilot study for treatment of jumper's knee. Injury. 2009 Jun;40(6):598-603. doi: 10.1016/j.injury.2008.11.026. Epub 2009 Apr 19. PMID 19380129
- [Background] Sanchez M, Anitua E, Azofra J, Andia I, Padilla S, Mujika I. Comparison of surgically repaired Achilles tendon tears using platelet-rich fibrin matrices. Am J Sports Med. 2007 Feb;35(2):245-51. doi: 10.1177/0363546506294078. Epub 2006 Nov 12. PMID 17099241
- [Background] Slater M, Patava J, Kingham K, Mason RS. Involvement of platelets in stimulating osteogenic activity. J Orthop Res. 1995 Sep;13(5):655-63. doi: 10.1002/jor.1100130504. PMID 7472743
- [Background] Peerbooms JC, Sluimer J, Bruijn DJ, Gosens T. Positive effect of an autologous platelet concentrate in lateral epicondylitis in a double-blind randomized controlled trial: platelet-rich plasma versus corticosteroid injection with a 1-year follow-up. Am J Sports Med. 2010 Feb;38(2):255-62. doi: 10.1177/0363546509355445. PMID 20448192
- [Background] Randelli P, Arrigoni P, Ragone V, Aliprandi A, Cabitza P. Platelet rich plasma in arthroscopic rotator cuff repair: a prospective RCT study, 2-year follow-up. J Shoulder Elbow Surg. 2011 Jun;20(4):518-28. doi: 10.1016/j.jse.2011.02.008. PMID 21570659
- [Background] Randelli PS, Arrigoni P, Cabitza P, Volpi P, Maffulli N. Autologous platelet rich plasma for arthroscopic rotator cuff repair. A pilot study. Disabil Rehabil. 2008;30(20-22):1584-9. doi: 10.1080/09638280801906081. PMID 18608363
- [Background] Mizuno H. Adipose-derived stem cells for tissue repair and regeneration: ten years of research and a literature review. J Nippon Med Sch. 2009 Apr;76(2):56-66. doi: 10.1272/jnms.76.56. PMID 19443990
- [Background] Casteilla L, Planat-Benard V, Laharrague P, Cousin B. Adipose-derived stromal cells: Their identity and uses in clinical trials, an update. World J Stem Cells. 2011 Apr 26;3(4):25-33. doi: 10.4252/wjsc.v3.i4.25. PMID 21607134
- [Background] Uysal AC, Mizuno H. Tendon regeneration and repair with adipose derived stem cells. Curr Stem Cell Res Ther. 2010 Jun;5(2):161-7. doi: 10.2174/157488810791268609. PMID 19941450
- [Background] Gimble J, Guilak F. Adipose-derived adult stem cells: isolation, characterization, and differentiation potential. Cytotherapy. 2003;5(5):362-9. doi: 10.1080/14653240310003026. PMID 14578098
- [Background] Zuk PA, Zhu M, Ashjian P, De Ugarte DA, Huang JI, Mizuno H, Alfonso ZC, Fraser JK, Benhaim P, Hedrick MH. Human adipose tissue is a source of multipotent stem cells. Mol Biol Cell. 2002 Dec;13(12):4279-95. doi: 10.1091/mbc.e02-02-0105. PMID 12475952
- [Background] Mizuno H, Hyakusoku H. Mesengenic potential and future clinical perspective of human processed lipoaspirate cells. J Nippon Med Sch. 2003 Aug;70(4):300-6. doi: 10.1272/jnms.70.300. PMID 12928709
- [Background] von Heimburg D, Hemmrich K, Haydarlioglu S, Staiger H, Pallua N. Comparison of viable cell yield from excised versus aspirated adipose tissue. Cells Tissues Organs. 2004;178(2):87-92. doi: 10.1159/000081719. PMID 15604532
- [Background] Smith RK, Webbon PM. Harnessing the stem cell for the treatment of tendon injuries: heralding a new dawn? Br J Sports Med. 2005 Sep;39(9):582-4. doi: 10.1136/bjsm.2005.015834. No abstract available. PMID 16118291
- [Background] Chong AK, Ang AD, Goh JC, Hui JH, Lim AY, Lee EH, Lim BH. Bone marrow-derived mesenchymal stem cells influence early tendon-healing in a rabbit achilles tendon model. J Bone Joint Surg Am. 2007 Jan;89(1):74-81. doi: 10.2106/JBJS.E.01396. PMID 17200313
- [Background] Ouyang HW, Goh JC, Thambyah A, Teoh SH, Lee EH. Knitted poly-lactide-co-glycolide scaffold loaded with bone marrow stromal cells in repair and regeneration of rabbit Achilles tendon. Tissue Eng. 2003 Jun;9(3):431-9. doi: 10.1089/107632703322066615. PMID 12857411
- [Background] Nixon AJ, Dahlgren LA, Haupt JL, Yeager AE, Ward DL. Effect of adipose-derived nucleated cell fractions on tendon repair in horses with collagenase-induced tendinitis. Am J Vet Res. 2008 Jul;69(7):928-37. doi: 10.2460/ajvr.69.7.928. PMID 18593247
- [Background] Gulotta LV, Kovacevic D, Ehteshami JR, Dagher E, Packer JD, Rodeo SA. Application of bone marrow-derived mesenchymal stem cells in a rotator cuff repair model. Am J Sports Med. 2009 Nov;37(11):2126-33. doi: 10.1177/0363546509339582. Epub 2009 Aug 14. PMID 19684297
- [Background] Del Bue M, Ricco S, Ramoni R, Conti V, Gnudi G, Grolli S. Equine adipose-tissue derived mesenchymal stem cells and platelet concentrates: their association in vitro and in vivo. Vet Res Commun. 2008 Sep;32 Suppl 1:S51-5. doi: 10.1007/s11259-008-9093-3. PMID 18683070
- [Background] Ellera Gomes JL, da Silva RC, Silla LM, Abreu MR, Pellanda R. Conventional rotator cuff repair complemented by the aid of mononuclear autologous stem cells. Knee Surg Sports Traumatol Arthrosc. 2012 Feb;20(2):373-7. doi: 10.1007/s00167-011-1607-9. Epub 2011 Jul 20. PMID 21773831
- [Background] MacIsaac ZM, Shang H, Agrawal H, Yang N, Parker A, Katz AJ. Long-term in-vivo tumorigenic assessment of human culture-expanded adipose stromal/stem cells. Exp Cell Res. 2012 Feb 15;318(4):416-23. doi: 10.1016/j.yexcr.2011.12.002. Epub 2011 Dec 13. PMID 22185824
- [Background] Guadalajara H, Herreros D, De-La-Quintana P, Trebol J, Garcia-Arranz M, Garcia-Olmo D. Long-term follow-up of patients undergoing adipose-derived adult stem cell administration to treat complex perianal fistulas. Int J Colorectal Dis. 2012 May;27(5):595-600. doi: 10.1007/s00384-011-1350-1. Epub 2011 Nov 9. PMID 22065114
- [Background] Guest DJ, Smith MR, Allen WR. Monitoring the fate of autologous and allogeneic mesenchymal progenitor cells injected into the superficial digital flexor tendon of horses: preliminary study. Equine Vet J. 2008 Mar;40(2):178-81. doi: 10.2746/042516408X276942. PMID 18267891
- [Background] Shiri R, Viikari-Juntura E, Varonen H, Heliovaara M. Prevalence and determinants of lateral and medial epicondylitis: a population study. Am J Epidemiol. 2006 Dec 1;164(11):1065-74. doi: 10.1093/aje/kwj325. Epub 2006 Sep 12. PMID 16968862
- [Background] Hohendorff B, Siepen W, Spiering L, Staub L, Schmuck T, Boss A. Long-term results after operatively treated Achilles tendon rupture: fibrin glue versus suture. J Foot Ankle Surg. 2008 Sep-Oct;47(5):392-9. doi: 10.1053/j.jfas.2008.05.006. Epub 2008 Jul 14. PMID 18725118
- [Background] Minagawa H, Yamamoto N, Abe H, Fukuda M, Seki N, Kikuchi K, Kijima H, Itoi E. Prevalence of symptomatic and asymptomatic rotator cuff tears in the general population: From mass-screening in one village. J Orthop. 2013 Feb 26;10(1):8-12. doi: 10.1016/j.jor.2013.01.008. eCollection 2013. PMID 24403741
- [Background] Jo CH, Shin JS, Lee YG, Shin WH, Kim H, Lee SY, Yoon KS, Shin S. Platelet-rich plasma for arthroscopic repair of large to massive rotator cuff tears: a randomized, single-blind, parallel-group trial. Am J Sports Med. 2013 Oct;41(10):2240-8. doi: 10.1177/0363546513497925. Epub 2013 Aug 6. PMID 23921338
- [Background] Oh JH, Chung SW, Kim SH, Chung JY, Kim JY. 2013 Neer Award: Effect of the adipose-derived stem cell for the improvement of fatty degeneration and rotator cuff healing in rabbit model. J Shoulder Elbow Surg. 2014 Apr;23(4):445-55. doi: 10.1016/j.jse.2013.07.054. Epub 2013 Oct 12. PMID 24129058
- [Background] Buchbinder R, Green SE, Struijs P. Tennis elbow. BMJ Clin Evid. 2008 May 28;2008:1117. PMID 19450309
- [Background] Levin D, Nazarian LN, Miller TT, O'Kane PL, Feld RI, Parker L, McShane JM. Lateral epicondylitis of the elbow: US findings. Radiology. 2005 Oct;237(1):230-4. doi: 10.1148/radiol.2371040784. Epub 2005 Aug 18. PMID 16118152
- [Derived] Chun SW, Kim W, Lee SY, Lim CY, Kim K, Kim JG, Park CH, Hong SH, Yoo HJ, Chung SG. A randomized controlled trial of stem cell injection for tendon tear. Sci Rep. 2022 Jan 17;12(1):818. doi: 10.1038/s41598-021-04656-z. PMID 35039529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment flyers were posted in a tertiary hospital and volunteers were recruited between September 2014 and April 2016. The first participant was enrolled on January 13, 2015 and the last participant was enrolled in April 12. 2016.
Pre-assignment Details: Volunteers were screened by a experienced physiatrist prior to enrollment. Of 26 potential participants, one refused to participate and another had incompatible findings in the baseline MRI. As a result, 24 participants met the inclusion/exclusion criteria and were enrolled and randomized to treatment.
Groups:
- Mesenchymal Stem Cell Group: Received allogenic adipose tissue-derived adult mesenchymal stem cells (10million cells) in fibrin glue scaffold.
  allogenic adipose stem cell injection: Intervention will be done with stem cell injection, 0.5cc (Total: 10 million cells), fibrin glue injection 0.5cc and range of motion exercise.
  Eight participants were assigned and one declined to participate before the intervention.
- Active Control (Fibrin Glue) Group: Received fibrin glue and normal saline.
  fibrin glue/normal saline injection: Total 1cc of fibin glue and normal saline mixture injection and range of motion exercise
  Eight participants were assigned and followed up throughout the study.
- Control (Normal Saline )Group: Received only normal saline.
  normal saline injection: Total 1cc of normal saline injection and range of motion exercise
  Eight participants were assigned and followed up throughout the study except one who missed the last visit.
Period: Overall Study
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
Started | 8 | 8 | 8
Intervention | 7 (Withdrawal by participant before intervention.) | 8 | 8
Completed | 7 | 8 | 8
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group | Total
Number analyzed (Participants) | 7 | 8 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (7.8) | 50.4 (4.6) | 54.1 (9.4) | 54.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 10
  Male | 3 | 4 | 6 | 13
Region of Enrollment [Number; unit: participants]
  South Korea | 7 | 8 | 8 | 23
Pain during activity [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale, scored from 0 to 10, higher score meaning worse outcome.
  units on a scale | 5.7 (1.6) | 4.7 (2.6) | 6.6 (2.4) | 5.7 (2.3)
Pain during rest [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale, scored from 0 to 10, higher score meaning worse outcome.
  units on a scale | 3.9 (1.8) | 2.4 (2.3) | 3.6 (1.8) | 3.3 (2.0)
American Shoulder and Elbow Surgeons (ASES) Shoulder Score [Mean (Standard Deviation); unit: units on a scale] — American Shoulder and Elbow Surgeons score, scored from 0 to 100, with higher scores indicating better outcomes
  units on a scale | 58.9 (12.1) | 64.7 (12.8) | 54.7 (20.1) | 59.5 (15.5)
University of California, Los Angeles(UCLA) Shoulder Score [Mean (Standard Deviation); unit: units on a scale] — University of California, Los Angeles(UCLA) Shoulder Score, range from 0 to 35 with a score of 0 indicating worse shoulder function and 35 indicating better shoulder function.
  units on a scale | 20.3 (3.7) | 19.0 (3.4) | 17.5 (3.0) | 17.9 (3.4)
The Disabilities of the Arm, Shoulder and Hand(DASH) Score [Mean (Standard Deviation); unit: units on a scale] — The Disabilities of the Arm, Shoulder and Hand(DASH) Score, scored 0 to 100, lower score meaning better outcome.
  units on a scale | 32.3 (13.0) | 35.2 (16.1) | 37.6 (23.8) | 35.1 (17.7)

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain During Activity From Baseline to 3 Months After Intervention
Description: Pain during activity will be evaluated by visual analog scale (active pain VAS). The active pain visual analog scale change from baseline to 3 months after intervention is the primary outcome. Visual analog scale is scored 0 to 10, higher scored meaning worse outcome. Negative values in change of pain during activity indicate improvement in pain.
Time Frame: Baseline and 3 months after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
Number analyzed (Participants) | 7 | 8 | 8
units on a scale | -1.4 (2.9) | -1.5 (2.4) | -3.0 (2.6)
Statistical Analysis 1: Comparison: Mesenchymal Stem Cell Group vs Active Control (Fibrin Glue) Group vs Control (Normal Saline )Group; Null hypothesis: There is no difference between the three groups. Statistical power: 0.80; Test type: Other; p = 0.35, Kruskal-Wallis

2. Secondary Outcome: Pain During Rest
Description: Pain during rest assessed by visual analog scale (VAS), scored 0 to 10, higher scores meaning worse outcome.
Time Frame: Baseline, 6 weeks, 12 weeks, 6, 12, 24 months after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
Number analyzed (Participants) | 7 | 8 | 8
units on a scale
  baseline | 3.9 (1.8) | 2.4 (2.3) | 3.6 (1.8)
  week 6 | 4.0 (2.1) | 2.2 (2.0) | 3.0 (1.7)
  month 3 | 2.8 (2.7) | 1.9 (1.7) | 2.7 (1.8)
  month 6 | 2.9 (1.9) | 1.4 (1.3) | 2.4 (2.1)
  month 12 | 2.9 (3.5) | 1.8 (2.4) | 1.3 (1.3)
  year 2 | 2.0 (2.2) | 0.8 (1.3) | 0.5 (0.8)
Statistical Analysis 1: Comparison: Mesenchymal Stem Cell Group vs Active Control (Fibrin Glue) Group vs Control (Normal Saline )Group; Test type: Equivalence — To test whether there were differences in the rate of change among groups; p = 0.662, Mixed Models Analysis

3. Secondary Outcome: Pain During Activity
Description: Pain during activity assessed by visual analog scale (VAS), scored 0 to 10, higher scores meaning worse outcome
Time Frame: Baseline, 6 weeks, 12 weeks, 6, 12, 24 months after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
Number analyzed (Participants) | 7 | 8 | 8
units on a scale
  baseline | 5.7 (1.6) | 4.7 (2.6) | 6.6 (2.4)
  week 6 | 6.0 (1.9) | 3.2 (2.1) | 4.6 (2.8)
  month 3 | 4.4 (2.9) | 3.2 (1.6) | 3.6 (2.0)
  month 6 | 4.3 (2.7) | 2.8 (2.3) | 4.3 (2.8)
  month 12 | 3.7 (2.7) | 3.2 (2.3) | 3.1 (2.4)
  year 2 | 4.4 (3.0) | 3.2 (2.1) | 1.1 (1.5)
Statistical Analysis 1: Comparison: Mesenchymal Stem Cell Group vs Active Control (Fibrin Glue) Group vs Control (Normal Saline )Group; Test type: Equivalence — To test whether there were differences in the rate of change among groups; p = 0.882, Mixed Models Analysis

4. Secondary Outcome: American Shoulder and Elbow Surgeons (ASES) Shoulder Score
Description: Functional score of the shoulder was assessed by American Shoulder and Elbow Surgeons shoulder score which is a questionnaire dedicated to the functional evaluation of the shoulder. It is scored from 0 to 100, higher scores meaning better outcome.
Time Frame: Baseline, 6 weeks, 12 weeks, 6, 12, 24 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
Number analyzed (Participants) | 7 | 8 | 8
score on a scale
  baseline | 58.9 (12.1) | 64.7 (12.8) | 54.7 (20.1)
  week 6 | 52.4 (21.0) | 70.6 (19.9) | 65.9 (15.8)
  month 3 | 67.9 (17.7) | 73.7 (15.3) | 63.6 (11.8)
  month 6 | 63.4 (19.6) | 76.7 (12.7) | 63.9 (14.9)
  month 12 | 70.6 (23.5) | 76.0 (20.3) | 74.4 (13.2)
  year 2 | 71.6 (20.3) | 80.0 (16.1) | 89.3 (11.5)
Statistical Analysis 1: Comparison: Mesenchymal Stem Cell Group vs Active Control (Fibrin Glue) Group vs Control (Normal Saline )Group; Test type: Equivalence — To test whether there were differences in the rate of change among groups; p = 0.835, Mixed Models Analysis

5. Secondary Outcome: Disability of Arm, Shoulder and Hand (DASH) Score
Description: Shoulder function is assessed by DASH score which is questionnaire dedicated to evaluate the function of the upper extremity. It is scored from 0 (no disability) to 100 (most severe disability).
Time Frame: Baseline, 6 weeks, 12 weeks, 6, 12, 24 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
Number analyzed (Participants) | 7 | 8 | 8
score on a scale
  baseline | 32.3 (13.0) | 35.2 (16.1) | 37.6 (23.8)
  week 6 | 36.7 (15.1) | 25.8 (16.9) | 28.1 (14.8)
  month 3 | 24.0 (15.0) | 19.2 (14.1) | 28.3 (10.7)
  month 6 | 25.0 (14.9) | 19.8 (11.1) | 27.1 (17.1)
  month 12 | 31.1 (20.8) | 20.5 (16.2) | 20.3 (13.7)
  year 2 | 20.3 (8.9) | 22.8 (16.8) | 20.1 (20.7)
Statistical Analysis 1: Comparison: Mesenchymal Stem Cell Group vs Control (Normal Saline )Group; Test type: Equivalence — To test whether there were differences in the rate of change among groups; p = 0.977, Mixed Models Analysis

6. Secondary Outcome: University of California, Los Angeles(UCLA) Shoulder Score
Description: Shoulder function is assessed by UCLA shoulder score which is a composite of range of motion examination and questionnaire dedicated to evaluate the function of the shoulder. It is scored from 0 to 35, higher scores meaning better shoulder function.
Time Frame: Baseline, 6 weeks, 12 weeks, 6, 12, 24 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
Number analyzed (Participants) | 7 | 8 | 8
score on a scale
  baseline | 20.3 (3.7) | 19.0 (3.4) | 17.5 (3.0)
  week 6 | 20.0 (6.4) | 22.3 (6.2) | 22.9 (5.9)
  month 3 | 26.4 (6.8) | 23.6 (6.0) | 21.4 (5.4)
  month 6 | 22.7 (6.5) | 23.6 (5.9) | 22.8 (4.9)
  month 12 | 23.6 (8.3) | 24.5 (7.2) | 28.0 (4.1)
  year 2 | 24.4 (6.7) | 24.6 (6.) | 31.3 (3.1)
Statistical Analysis 1: Comparison: Mesenchymal Stem Cell Group vs Active Control (Fibrin Glue) Group vs Control (Normal Saline )Group; Test type: Equivalence — To test whether there were differences in the rate of change among groups; p = 0.867, Mixed Models Analysis

7. Secondary Outcome: Tear Size at 3 Months After Injection
Description: Tear size was evaluated by 3-point Likert scale using MRI. The 3months follow-up images were compared to the baseline image and graded either; improved, stationary, and aggravated.
Time Frame: baseline and 3 months after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
Number analyzed (Participants) | 7 | 8 | 8
Participants
  stationary at month 3 | 5 | 5 | 5
  improved at month 3 | 2 | 2 | 2
  aggravated at month 3 | 0 | 1 | 1
Statistical Analysis 1: Comparison: Mesenchymal Stem Cell Group vs Active Control (Fibrin Glue) Group vs Control (Normal Saline )Group; Test type: Equivalence — To test whether there were differences in the change of tear size among groups; p = 0.916, Chi-squared

8. Secondary Outcome: Tear Size at 12 Months After Injection
Description: Tear size was evaluated by 3-point Likert scale using MRI. The 12 months follow-up images were compared to the baseline image and graded either; improved, stationary, and aggravated.
Time Frame: baseline and12 months after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
Number analyzed (Participants) | 7 | 8 | 8
Participants
  stationary at month 12 | 4 | 3 | 4
  improved at month 12 | 1 | 3 | 2
  aggravated at month 12 | 2 | 2 | 2
Statistical Analysis 1: Comparison: Mesenchymal Stem Cell Group vs Active Control (Fibrin Glue) Group vs Control (Normal Saline )Group; Test type: Equivalence — To test whether there were differences in the change of tear size among groups; p = 0.892, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 years
Description: All participants were asked the following open questions at every follow-up visit.
  1. How are you feeling?
  2. Have you had any kind of medical issue since the last visit?
  3. Have you had or currently on any medication since the last visit?
  4. Have you visited the emergency room or have been admitted to a hospital since the last visit?
Arm/Group | Mesenchymal Stem Cell Group | Active Control (Fibrin Glue) Group | Control (Normal Saline )Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesenchymal Stem Cell Group (N=7) | Active Control (Fibrin Glue) Group (N=8) | Control (Normal Saline )Group (N=8)
insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (11) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No